CLINICAL TRIAL: NCT02004574
Title: Investigator Initiated Study for Optimal Maintenance Treatment With Calcipotriol /Betamethasone Dipropionate Gel in Korean Patients With Psoriasis Vulgaris
Brief Title: Study for Treatment With Calcipotriol/Betamethasone Dipropionate Gel in Korean Patients With Psoriasis Vulgaris
Acronym: TRIANGLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jooheung Lee (Other)
Responsible Party: Sponsor-Investigator, Jooheung Lee, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSPLK 2013-01
Record Dates: First submitted 2013-11-10; First posted 2013-12-09 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene; betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PRN treatment (Experimental): Group 1: PRN treatment Apply Xamiol® gel (Calcipotriol/betamethasone dipropionate gel) once daily as needed (PRN)
  Interventions: Drug: Calcipotriol/betamethasone dipropionate gel
- Continuous treatment (Experimental): Group 2: Continuous treatment Apply Xamiol® gel (Calcipotriol/betamethasone dipropionate gel)once daily
  Interventions: Drug: Calcipotriol/betamethasone dipropionate gel
- Weekends treatment (Experimental): Group 3: Weekends treatment (twice weekly) Apply Xamiol® gel (Calcipotriol/betamethasone dipropionate gel) once daily at weekends (on Saturdays and Sundays)
  Interventions: Drug: Calcipotriol/betamethasone dipropionate gel

INTERVENTIONS:
Drug: Calcipotriol/betamethasone dipropionate gel — All enrolled subjects will receive Xamiol® gel once daily for 8 weeks during the induction period and then will be assessed according to IGA at the end of 8-week induction period. Those subjects determined to be "Responder" by IGA will be randomized to one of the following three treatment groups and they will continue their therapy with randomized maintenance regimens for the duration of additional 8 weeks.
  Other Names: Xamiol gel

SUMMARY:
The combination of calcipotriol and betamethasone dipropionate used in an ointment formulation (Daivobet® ointment) has shown to have an excellent efficacy and safety in the short-term and long-term management of psoriasis vulgaris. A newly developed gel formulation (Xamiol® gel) of calcipotriol and betamethasone dipropionate has recently been approved and marketed in Korea as a topical treatment of moderate to severe scalp psoriasis and non-scalp psoriasis vulgaris.

Xamiol® gel, the investigational product (IP) used in this study, prevents keratinization by normalizing the reproduction cycle of skin cells. It also relieves itching associated with psoriasis. Xamiol® gel was initially approved for treatment of moderate to severe scalp psoriasis and its label was extended to non-scalp psoriasis vulgaris in October 2012.

Since patient compliance is one of the important factors in achieving effective outcomes in the treatment of psoriasis, the once daily dosing of Xamiol® gel is expected to enhance compliance and treatment outcomes as well as to provide a safe and effective therapeutic option.

DETAILED DESCRIPTION:
Psoriasis is a disease difficult to cure and is usually recurrent and therefore, a continued management is crucial. An evidence-based approach is important for appropriate treatments of patient with psoriasis. However, there is a lack of response data for the topical treatments in Asian patients with psoriasis, and no treatment guidelines available. Therefore, routine topical treatments, instead of patient-specific treatments, are usually applied, which may result in treatment failure. In this regard, it is imperative to conduct a study to assess topical treatments in Korean patients with psoriasis vulgaris in terms of efficacy and side effects.

Furthermore, psoriasis patients in Korea, mostly small plaque types, may exhibit different disease activities and response outcomes and accordingly require different treatment options as compared to Western populations whose dominant psoriasis type is large plaque type. Thus, a study in Korean patients with psoriasis may reveal an interesting finding.

In order to investigate optimal maintenance regimens for the topical treatment of Korean patients with psoriasis vulgaris, we are planning this study which evaluates the efficacy of three 8-week maintenance regimens containing Xamiol® gel (PRN treatment group, Continuous treatment group and Twice weekly treatment group) in patients who have become "Responder" after 8-week induction therapy with Xamiol® gel ("Responder").

The primary objective of this study is to evaluate the percentages of "Responder"* at week 16, as assessed by Investigator's Global Assessment of Disease Severity (IGA), in three different 8-week maintenance regimens of Xamiol® gel after 8-week induction treatment with Xamiol® gel in patients with psoriasis vulgaris.

* Responder is defined as subjects with "clear" or "almost clear" according to IGA.

Secondary study objectives is to evaluate efficacy, % of Relapse and time to Relapse, PGA, Patient Compliance, Safety and Quality of Life (DLQI and TSQM) in three arms with calcipotriol/betamethasone dipropionate combination gel treatment in Korean patients with chronic plaque psoriasis of the body.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 19 years and above
2. Clinical diagnosis of stable psoriasis vulgaris of at least 4 weeks duration involving the non-scalp regions of the body (trunk and/or limbs) amenable to treatment with a maximum of 100 g of topical medication per week at screening
3. An investigator's global assessment of disease severity(IGA) of at least mild on the body (trunk and/or limbs) at Day 0 (Baseline)
4. Signed written informed consent prior to performance of any study-specific procedures or assessments, and must be willing to comply with treatment and follow up
5. Able to communicate with the investigator and understand and comply with the requirements of the study
6. Women of childbearing potential must have a negative pregnancy test and must use adequate contraception during the treatment phase of the study and for at least 1 week after the last application of study medication

Exclusion Criteria:

1. Body surface area (BSA) > 10 % or Psoriasis Area and Severity Index (PASI) > 10 at baseline

   * The palm of one hand is approximately 1 percent of the body surface area
2. Subjects with unstable forms of psoriasis including guttate, erythrodermic, exfoliative and pustular psoriasis, or psoriatic arthritis
3. Subjects with known disorders of calcium metabolism/hypercalcemia
4. Subjects with hypersensitivity to the active substances or to any of the excipients of the investigational products
5. Systemic treatment with biological therapies with a possible effect on psoriasis vulgaris within the following time periods prior to baseline visit

   * etanercept - within 4 weeks prior to baseline
   * adalimumab, alefacept, infliximab - within 2 months prior to baseline
   * ustekinumab - within 4 months prior to baseline
   * investigational product - within 4 weeks/5 half-lives (whichever is longer) prior to baseline
6. Systemic treatment with all other therapies with a possible effect on psoriasis vulgaris (e.g., corticosteroids, retinoids, methotrexate, cyclosporine and other immunosuppressants) within 4 weeks prior to baseline visit
7. Phototherapy within the following time periods prior to baseline visit

   * PUVA or Grenz ray - within 4 weeks
   * UV-B - within 2 weeks
8. Any topical treatment of the trunk and/or limbs (except for emollients) within 2 weeks prior to baseline visit
9. Topical treatment for other relevant skin disorders on the face and flexures (e.g., facial and flexural psoriasis, eczema) with class 1- 5 corticosteroids or vitamin D analogues within 2 weeks prior to baseline visit
10. Topical treatment for other relevant skin disorders on the scalp (e.g. scalp psoriasis) with class 1-5 corticosteroids, vitamin D analogues within 2 weeks prior to baseline visit
11. Subjects with severe renal insufficiency
12. Subjects with severe hepatic disorders
13. Subjects with a confounding skin condition or disorders against psoriasis evaluation
14. Subjects with viral (e.g. herpes or varicella) lesions of the skin, fungal or bacterial skin infections, parasitic infections on the treatment area
15. Subjects with skin manifestations in relation to tuberculosis or syphilis on the treatment area
16. Subjects with perioral dermatitis, atrophic skin, striae atrophicae on the treatment area
17. Subjects with fragility of skin veins, ichthyosis on the treatment area
18. Subjects with acne vulgaris, rosacea, wounds, ulcers, perianal and genital pruritus on the treatment area
19. Planned initiation of, or changes to, concomitant medication that could affect psoriasis vulgaris (e.g. beta blockers, anti-malarials, lithium, ACE inhibitors) during the study
20. Pregnant or lactating female subjects
21. Subjects who are planning a pregnancy during the entire study period

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Percentage of "Responder" (subjects with a grade of "clear" or "almost clear") according to IGA at Week 16 | Week 16
  The primary objective of this study is to evaluate the percentages of "Responder"* at week 16, as assessed by Investigator's Global Assessment of Disease Severity (IGA), in three different 8-week maintenance regimens of Xamiol® gel after 8-week induction treatment with Xamiol® gel in patients with psoriasis vulgaris.

SECONDARY OUTCOMES:
Investigator's global assessment of disease severity | Week 0, 4, 8, 12 and 16
  To evaluate the change of disease severity assessed by IGA in induction treatment phase and compare the IGA disease severity of three different maintenance regimens in the maintenance treatment phase.
Percentage of disease relapse | Week 0, 4, 8, 12 and 16
  To evaluate descriptive statistics of three different regimens in the maintenance treatment phase and compare percentage of relapse in threee different regimens.
Patient's global assessment of disease severity | Week 0, 4, 8, 12 and 16
  To evaluate the change of disease severity assessed by PGA in induction treatment phase and compare the PGA disease severity of three different maintenance regimens in the maintenance treatment phase.
Change in Psoriasis Area and Severity Index (PASI) score from Baseline to Week | Week 0, 4, 8, 12 and 16
  To evaluate the change of PASI in induction treatment phase and compare the PASI of three different maintenance regimens in the maintenance treatment phase.
Percent of subjects achieving a 75% improvement in the Psoriasis Area and Severity Index (PASI) score | Week 0, 4, 8, 12 and 16
  To evaluate the change of PASI75 from week 4 to week 8 in induction treatment phase and compare PASI75 in three different regimens in the maintenance treatment phase.
Time to relapse | Week 0, 4, 8, 12 and 16
  To evaluate descriptive statistics of three different regimens in the maintenance treatment phase and compare the time to relapse in threee different regimens.

OTHER OUTCOMES:
Subject's Compliance | Week 4, 8, 12 and 16
  To evaluate subject's compliance by subject's diary, interview, used IP dose and evaluate descriptive statistics for them.
Dermatology Life Quality Index | Week 0, 4, 8, 12 and 16
  To evaluate the change of DLQI score in induction treatment phase and evaluate change rate of week 8, week 12 and week 16 compared with baseline in the maintenance treatment phase.
Treatment Satisfaction Questionnaire for Medication | Week 8 and 16
  To evaluated descriptive statistics for TSQM score of week 8 in the induction treatment phase and evaluate change rate of week 8, week 16 and from week 8 to week 16 in the maintenance treatment phase.
Other treatment after completion of study | Week 16
  To evaluate descriptive statistics for used other medication after study completion.
Laboratory assessment | Week 0, 8, 16 and 18
  To evaluate the reported values(normal/abnormal) as follows.
  : To evaluate change of reported values from baseline to week 8 in induction treatment phase and compare reported values of week 8 and week 16 in three different regimens in the maintenance treatment phase.
SAEs | Week 0, 4, 8, 12, 16 and 18
  To evaluate the number of occurrance(subject-based) in each treatment phase and regimen and compare the number of occurrance in three difference regimens in the maintenance treatment phase.
AEs | Week 0, 4, 8, 12, 16 and 18
  To evaluate the number of occurrance(subject-based) in each treatment phase and regimen and compare the number of occurrance in three difference regimens in the maintenance treatment phase.
ADRs | Week 0, 4, 8, 12, 16 and 18
  To evaluate the number of occurrance(subject-based) in each treatment phase and regimen and compare the number of occurrance in three difference regimens in the maintenance treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Heung Lee, MD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Gangnam-gu, Seoul, South Korea

REFERENCES:
- [Result] Lowes MA, Bowcock AM, Krueger JG. Pathogenesis and therapy of psoriasis. Nature. 2007 Feb 22;445(7130):866-73. doi: 10.1038/nature05663. PMID 17314973
- [Result] Lew W, Lee E, Krueger JG. Psoriasis genomics: analysis of proinflammatory (type 1) gene expression in large plaque (Western) and small plaque (Asian) psoriasis vulgaris. Br J Dermatol. 2004 Apr;150(4):668-76. doi: 10.1111/j.0007-0963.2004.05891.x. PMID 15099362
- [Result] Pariser DM, Bagel J, Gelfand JM, Korman NJ, Ritchlin CT, Strober BE, Van Voorhees AS, Young M, Rittenberg S, Lebwohl MG, Horn EJ; National Psoriasis Foundation. National Psoriasis Foundation clinical consensus on disease severity. Arch Dermatol. 2007 Feb;143(2):239-42. doi: 10.1001/archderm.143.2.239. PMID 17310004
- [Result] Kragballe K, Austad J, Barnes L, Bibby A, de la Brassinne M, Cambazard F, Fleming C, Heikkila H, Williams Z, Peyri Rey J, Svensson A, Toole J, Wozel G. Efficacy results of a 52-week, randomised, double-blind, safety study of a calcipotriol/betamethasone dipropionate two-compound product (Daivobet/Dovobet/Taclonex) in the treatment of psoriasis vulgaris. Dermatology. 2006;213(4):319-26. doi: 10.1159/000096069. PMID 17135738
- [Result] Kragballe K, Noerrelund KL, Lui H, Ortonne JP, Wozel G, Uurasmaa T, Fleming C, Estebaranz JL, Hanssen LI, Persson LM. Efficacy of once-daily treatment regimens with calcipotriol/betamethasone dipropionate ointment and calcipotriol ointment in psoriasis vulgaris. Br J Dermatol. 2004 Jun;150(6):1167-73. doi: 10.1111/j.1365-2133.2004.05986.x. PMID 15214905
- [Result] Langley RG, Gupta A, Papp K, Wexler D, Osterdal ML, Curcic D. Calcipotriol plus betamethasone dipropionate gel compared with tacalcitol ointment and the gel vehicle alone in patients with psoriasis vulgaris: a randomized, controlled clinical trial. Dermatology. 2011;222(2):148-56. doi: 10.1159/000323408. Epub 2011 Feb 3. PMID 21293107
- [Result] Samarasekera E, Sawyer L, Parnham J, Smith CH; Guideline Development Group. Assessment and management of psoriasis: summary of NICE guidance. BMJ. 2012 Oct 24;345:e6712. doi: 10.1136/bmj.e6712. No abstract available. PMID 23097521